CLINICAL TRIAL: NCT06321861
Title: The Effects of Caffeine Supplementation on Motivation, Affect and Performance in Physical Exercise Tests: An Intervention Study
Brief Title: Motivational, Affective and Performance Effects of Caffeine Supplementation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Collaborators: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other); University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Principal Investigator, Ewa Szumowska, Assistant, Jagiellonian University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Caffeine_motivation
Record Dates: First submitted 2024-01-17; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Caffeine; Affect; Goals
Keywords: caffeine; energization; motivation; effort; affect; physical exercise; arousal
MeSH Terms: conditions — Motor Activity | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: Each participant will take part in three similar sessions differing by the substance they receive: caffeine (intervention group), placebo, no substance. Sessions will be about one week apart.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caffeine (Experimental): Participants will take a caffeine pill (3mg/kg of body mass) 60 minutes before the physical exercise test.
  Interventions: Dietary Supplement: Caffeine
- Placebo (Placebo Comparator): Participants will take a placebo pill 60 minutes before the physical exercise test.
  Interventions: Dietary Supplement: Placebo
- No substance (Other): Participants receive no pills in this condition before the physical exercise test.
  Interventions: Other: No substance

INTERVENTIONS:
Dietary Supplement: Caffeine — Participants will take one caffeine pill. The dose of caffeine will be calculated based on participants' body mass (3mg/kg body mass). Caffeine will be provided in capsules containing the individual amount of caffeine and will be administered orally 60 min before the onset of the exercise protocol.
  Arms: Caffeine
Dietary Supplement: Placebo — Participants will take one pill with no caffeine in it. The manufacturer of the caffeine capsules will also prepare identical placebo capsules filled out with a microcrystalline cellulose. Placebo will be administered orally 60 min before the onset of the exercise protocol.
  Arms: Placebo
Other: No substance — Participants will take no substance. They will just wait 60 minutes and then engage in the exercise protocol.
  Arms: No substance

SUMMARY:
The main objective of the study is to evaluate the influence of caffeine intake on participants' energetic arousal, affect, motivation to achieve a training goal, satisfaction with training, and the sense of agency during training. Consequently, participants will engage in three sessions: caffeine, placebo, and no substance (in counterbalanced order). During each session, their affective and motivational states will be assessed, along with the performance of a standardized physical exercise test. The investigators hypothesize that participants who consume caffeine (caffeine condition) will exhibit higher levels of energy and motivation compared to the other two groups. Additionally, they are expected to experience greater optimism and expectancy regarding their training goals and achieve better results in the physical exercise test.

A secondary aim of the study is to examine the impact of genetic variability on motivational and affective states of participants, as well as their performance in the physical exercise test after caffeine. The investigators will assess the CYP1A2 (-163C > A, rs762551; characterized such as "fast" (AA genotype) and "slow" caffeine metabolizers (C-carriers)) and ADORA2A (1976T > C; rs5751876; characterized by "high" (TT genotype) or "low" sensitivity to caffeine (C-carriers)).

DETAILED DESCRIPTION:
Before participating in the study, participants will answer questions regarding their consumption of caffeinated beverages and the frequency of their workouts. They will also complete the Extreme Personality Scale measuring the tendency to pursue goals single-mindedly. Subsequently, they will be qualified for the study based on the questionnaire results and a brief interview.

The study will involve the manipulation of energization through the administration of caffeine. Participants will take part in a randomized, crossover, double-blind study, where they will perform three identical training sessions after consuming: a) caffeine at a dose of 3 mg/kg of body weight; b) a placebo; and c) under control conditions (i.e., without substance administration). Capsule consumption will occur 60 minutes before the start of the training. Caffeine and placebo capsules will not differ in size, shape, color, and taste.

As the effectiveness of caffeine use depends on the CYP1A2 (rs762551) and ADORA2 (rs5751876) gene polymorphisms, the study will also genotype these genes. The first gene is responsible for the rate of caffeine metabolism, determining whether people metabolize caffeine "fast" or "slow." The ADORA2A gene, encoding the adenosine A2A receptor, influences how "sensitive" people are to caffeine. DNA isolates obtained from oral epithelial cells collected from participants by qualified medical personnel will constitute the research material. Oral epithelial swabs will be collected directly from the participants into sterile tubes.

Before and after substance intake (and additionally after the exercise test) participants will assess their arousal using the University of Wales Institute of Science and Technology Mood Adjective Checklist. Additionally, after substance intake and before exercise, participants will answer questions about motivation, affect and expectancy regarding training. Subsequently, participants will undergo training, taking the form of a supervised standardized exercise test. After exercise, participants will assess their satisfaction and feelings after completing the training.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years
* Caffeine consumption
* Engagement in physical activity.

Exclusion Criteria:

* Diagnosed cardiovascular, metabolic, gastrointestinal, or neurological diseases
* Taking medications or supplements that may affect test results
* Tobacco smoking
* Pregnancy
* Potential allergy to caffeine.

Participation in the study will be preceded by completing a health questionnaire and providing written consent. Additionally, exclusion from the study will occur upon the explicit request of the participant.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Energetic arousal pre-test | Right before the intervention
  Self-reported energetic arousal contrasting vigour with fatigue, measured with the energetic arousal sub-scale of the University of Wales Institute of Science and Technology Mood Adjective Checklist. The values range from 1-4; higher scores indicate greater energetic arousal.
Energetic arousal post-test | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Self-reported energetic arousal measured with the energetic arousal sub-scale of the University of Wales Institute of Science and Technology Mood Adjective Checklist. The values range from 1-4; higher scores indicate greater energetic arousal. The change relative to the pre-test will be analyzed.
Optimism | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Situational optimism (expectancy of positive outcomes) measured with 4 items were participants rate the extent to which they: 1) are positively oriented. 2) are full of optimism. 3) can achieve what I set out to do. 4) are capable of a lot. Responses are given on a 1-7 Likert scale. Higher scores indicate greater optimism. The mean of these items will be computed and the change relative to the pre-test will be analyzed.
Motivation | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Motivation to accomplish one's training goals measured with a question where participants rate the extent to which they are motivated to achieve the best result in: 1) one-repetition maximum bench press test, 2) bar velocity in the bench press test, 3) strength-endurance test, 4) countermovement jump. Participants respond to each item on a 1-7 Likert scale. Higher scores indicate greater motivation.
Determination | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Determination to accomplish one's training goals measured with 4 items: 1) During training, everything else will become irrelevant for [the participant[. 2) [The participant] will put a lot of energy into the training. 3) [The participant] will do everything in their power to achieve the training goal. 4) [The participant] will reach the training goal even if it requires a great effort. 5) [The participant] will train despite fatigue. Participants respond to each item on a 1-7 Likert scale. Higher scores indicate greater determination.
Relative outcome expectancy | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Expectancy of the training results measured with a question: In relation to participants' typical result, what result do they expect in: 1) one-repetition maximum bench press test, 2) bar velocity in the bench press test, 3) strength-endurance test, 4) countermovement jump. Participants respond to each item on a 1-7 scale anchored 1 = definitely worse than usual and 7 = definitely better than usual. Higher scores indicate more positive outcome expectations.
Success probability | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Subjective probability of attaining the best result measured with a question: How likely do participants think it is that they will achieve the best result in: 1) one-repetition maximum bench press test, 2) bar velocity in the bench press test, 3) strength-endurance test, 4) countermovement jump. Participants respond to each item on a 1-7 scale anchored 1 = completely unlikely and 7 = certain. Higher scores indicate greater probability of success.
Prospective effort | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Participants' willingness to invest effort in the training measured with a question: How much effort are participants planning to invest in: 1) one-repetition maximum bench press test, 2) bar velocity in the bench press test, 3) strength-endurance test, 4) countermovement jump. Participants respond on a 0-100% scale. Higher scores indicate greater willingness to invest effort.
Agency | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Sense of agency measured with two questions: 1) Do participants feel in control over the outcome in..., 2) Do participants feel in control over their performance in... Participants respond to each question in relation to each test outcome: 1) one-repetition maximum bench press test, 2) bar velocity in the bench press test, 3) strength-endurance test, 4) countermovement jump. Responses are given on 1-6 scale anchored 1 = no control and 7 = complete control. Higher scores indicate greater sense of agency.
Performance in the 1RM test | 60 minutes after taking the capsule (waiting in the no-intervention condition)
  Participants' performance in the one-repetition maximum test in bench press [number of kg]
Performance in the bar velocity in the bench press test | 60 minutes after taking the capsule (waiting in the no-intervention condition)
  Participants' performance in the bar velocity during 3 sets of 3 repetitions in the bench press exercise [m/s]
Performance in the strength-endurance test | 60 minutes after taking the capsule (waiting in the no-intervention condition)
  Participants' performance in the strength-endurance test in bench press test (number of repetitions)
Performance in the countermovement jump test | 60 minutes after taking the capsule (waiting in the no-intervention condition)
  Participants' performance in the countermovement jump test (number of cm)
Satisfaction with the results | Immediately after the physical exercise test
  Participants' satisfaction with their training results measured with a question: How satisfied are participants with their results in: 1) one-repetition maximum bench press test, 2) bar velocity in the bench press test, 3) strength-endurance test, 4) countermovement jump. Participants respond to each item on a 1-7 scale anchored 1 = definitely unsatisfied to 7 = definitely satisfied. Higher scores indicate greater satisfaction with the results.
Retrospective effort | Immediately after the physical exercise test
  Participants' assessment of effort invested in the training measured with a question: How much effort did participants invest in:1) one-repetition maximum bench press test, 2) bar velocity in the bench press test, 3) strength-endurance test, 4) countermovement jump. Participants respond on a 0-100% scale. Higher scores indicate greater effort.
Retrospective agency | Immediately after the physical exercise test
  Sense of agency measured with two questions: 1) Did participants feel in control over the outcome in..., 2) Did participants feel in control over their performance in... Participants respond to each question in relation to each test outcome: 1) one-repetition maximum bench press test, 2) bar velocity in the bench press test, 3) strength-endurance test, 4) countermovement jump. Responses are given on 1-6 scale anchored 1 = no control and 7 = complete control. Higher scores indicate greater sense of agency.

SECONDARY OUTCOMES:
Goal importance | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Importance of the training goal measured with a question: How important is it for participants to achieve the best possible result in: 1) one-repetition maximum bench press test, 2) bar velocity in the bench press test, 3) strength-endurance test, 4) countermovement jump. Participants respond to each item on a 1-7 scale anchored 1 = completely unimportant and 7 = extremely important. Higher scores indicate greater importance.
Prospective difficulty | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Perceived difficulty of the training goal measured with a question: How do participants assess the difficulty of: 1) one-repetition maximum bench press test, 2) bar velocity in the bench press test, 3) strength-endurance test, 4) countermovement jump. Participants respond to each item on a 1-7 scale anchored 1 = definitely easy and 7 = definitely difficult. Higher scores indicate greater subjective difficulty.
Expected performance in the 1RM test | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Participants' expected performance in the 1 RM test. Participants provide responses to the following questions:
  How much weight do participants think they will lift in the 1 RM test? (participants provide in kg)
Expected performance in the bar velocity in the bench press test | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Participants' expected performance in the bar velocity in the bench press test. Participants provide a response to the following question:
  How much m/s. do participants expect to achieve in the bar velocity test? (participants provide the response in m/s)
Expected performance in the strength-endurance test | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Participants' expected performance in the strength-endurance test. Participants provide a response to the following question:
  How many repetitions do participants think they will perform in the strength-endurance test? (participants provide the number of repetitions)
Expected performance in the countermovement jump test | 60 minutes after taking the capsule (waiting in the no-intervention condition); before training
  Participants' expected performance in the countermovement jump test. Participants provide a response to the following question:
  How high do participants think they will jump? (participants provide in cm)
Retrospective difficulty | Immediately after the physical exercise test
  Assessed difficulty of each training element: 1) one-repetition maximum bench press test, 2) bar velocity in the bench press test, 3) strength-endurance test, 4) countermovement jump. Participants rate each element twice (generally and in relation to their other trainings) on a 1-7 scale anchored 1 = very easy and 7 = very difficult. Higher scores indicate greater difficulty.
Energetic arousal post-training | Immediately after the physical exercise test
  Self-reported energetic arousal measured with the energetic arousal sub-scale of the University of Wales Institute of Science and Technology Mood Adjective Checklist. The values range from 1-4; higher scores indicate greater energetic arousal.
Perceived effect on agency | Immediately after the physical exercise test
  Assessed effect on the sense of agency measured with an item:
  To what extent do participants agree with the statement: Completing this workout made participants feel like they had control. Participants respond on 1-7 Likert scale. Higher scores indicate the greater perceived effect on agency.
Tense arousal | Right before the intervention, then 60 minutes after taking the capsule (waiting in the no-intervention condition); and immediately after the physical exercise test
  Self-reported tense arousal contrasting tension with relaxation, measured with the Tense Arousal subscale of the University of Wales Institute of Science and Technology Mood Adjective Checklist. The values range from 1-4; higher scores indicate greater energetic arousal.
Hedonic tone | Right before the intervention, then 60 minutes after taking the capsule (waiting in the no-intervention condition); and immediately after the physical exercise test
  Self-reported hedonic tone contrasting pleasant with unpleasant moods, measured with the Hedonic Tone subscale of the University of Wales Institute of Science and Technology Mood Adjective Checklist. The values range from 1-4; higher scores indicate greater energetic arousal.

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Szumowska, Principal Investigator — Jagiellonian University
Locations (1):
- The Jerzy Kukuczka Academy of Physical Education in Katowice, Katowice, Poland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD will be shared digitally via the Jagiellonian University Repository.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: The data will become available after preparing the article summarizing the study results. The data will be shared for at least 5 years.
Access Criteria: All researchers possessing the link to the data will be able to access it.

REFERENCES:
- [Background] Matthews G; Jones DM, Chamberlain AG. Refining the measurement of mood: The UWIST mood adjective checklist. British Journal of Psychology, 1990, 81(1): 17-42.
- [Background] Szumowska E, Molinario E, Jaśko K, Hudiyana J, Firdiani NF, Penrod J, Jaume LC, Leander NP, Kreienkamp J, Agostini M, Gruszka A, Szumska I, Stelmaszyńska D, Gola M, Altungy P, Gómez Á, Cacek J, & Kruglanski AW (2023). The Extreme Personality: Individual Differences in Proneness to Motivational Imbalance. Manuscript submitted for publication.